CLINICAL TRIAL: NCT04803747
Title: A Phase IV Trial of a Hospital Policy of Tranexamic Acid Use to Reduce Transfusion in Major Non-cardiac Surgery (TRACTION): A Pragmatic Randomized Cluster Crossover Trial
Brief Title: A Trial of a Hospital Policy of Tranexamic Acid Use to Reduce Transfusion in Major Non-cardiac Surgery
Acronym: TRACTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Sciences Centre Foundation, Manitoba (Other); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ryan Zarychanski, Nominated Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TXA-51231
Record Dates: First submitted 2021-02-01; First posted 2021-03-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Major Non-cardiac Surgeries
Keywords: Tranexamic acid (TXA); Venous thromboembolism (VTE); Deep vein thrombosis (DVT); Transfusion; Perioperative Bleeding
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: TRACTION is a pragmatic, multicenter, randomized, registry-based cluster-crossover trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Over the duration of the study, participating centres will be centrally and randomly allocated to receive either TXA or matching placebo at 1-month intervals for a total of 8 months. Intervention assignment will only be known to the research pharmacy staff who will prepare the study drug specific to the interval assignment. To minimize sources of selection and ascertainment biases, anesthesiologists, surgeons, investigators, research staff, and members of the Data Safety and Monitoring Board will all be blinded to randomization schemes and treatments administered; only the trial statistician will have access to randomization schemes for all sites. The research site's Pharmacy staff will not have contact with the study team or the patient and will be expressly forbidden to discuss individual treatment allocation with the study team, the patient, the operating room and clinical care team unless emergency un-blinding is warranted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (TXA) Arm (Active Comparator): TXA 1 gram bolus (2 grams for patients over 100 kg) intravenously (IV) administered within 10 minutes of the first surgical incision, followed by 1 additional gram given intravenously at 2-4 hours of surgery or prior to skin closure, at the discretion of the anesthesiologist (e.g. IV bolus at 2-4 hours of surgery, at skin closure, or the 1 additional gram given as a continuous infusion throughout the surgical procedure).
  Interventions: Drug: Tranexamic acid (TXA)
- Placebo Arm (Placebo Comparator): Placebo 1 gram bolus (2 grams for patients over 100 kg) intravenously (IV) administered within 10 minutes of the first surgical incision, followed by 1 additional gram given intravenously at 2-4 hours of surgery or prior to skin closure, at the discretion of the anesthesiologist (e.g. IV bolus at 2-4 hours of surgery, at skin closure, or the 1 additional gram given as a continuous infusion throughout the surgical procedure).
  Interventions: Drug: Placebo (0.9 % Saline)

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — TXA 1 gram bolus (2 grams for patients over 100 kg) intravenously (IV) administered within 10 minutes of the first surgical incision, followed by 1 additional gram given intravenously at 2-4 hours of surgery or prior to skin closure, at the discretion of the anesthesiologist (e.g. IV bolus at 2-4 hours of surgery, at skin closure, or the 1 additional gram given as a continuous infusion throughout the surgical procedure).
  Arms: Tranexamic acid (TXA) Arm
Drug: Placebo (0.9 % Saline) — Placebo (0.9 % normal saline) 1 gram bolus (2 grams for patients over 100 kg) intravenously (IV) administered within 10 minutes of the first surgical incision, followed by 1 additional gram given intravenously at 2-4 hours of surgery or prior to skin closure, at the discretion of the anesthesiologist (e.g. IV bolus at 2-4 hours of surgery, at skin closure, or the 1 additional gram given as a continuous infusion throughout the surgical procedure).
  Arms: Placebo Arm

SUMMARY:
A Phase IV trial of a hospital policy of Tranexamic acid to reduce transfusion in major non-cardiac surgery.

DETAILED DESCRIPTION:
The TRACTION Trial is a national multi-centre Phase IV randomized cluster-crossover trial of Tranexamic acid versus placebo. Over the duration of the study, participating centres will be centrally and randomly allocated to receive either TXA or matching placebo at 1-month intervals. As our pragmatic trial is designed to define practice, we have selected co-primary outcomes that evaluate effectiveness in the context of safety.

Our co-primary outcomes are the:

1. Proportion of patients transfused RBCs
2. Incidence of DVT or PE (collectively called venous thromboembolism (VTE) within 90 days of surgery.

ELIGIBILITY:
Cluster-level inclusion criteria:

Hospital sites will be included in the trial if the site performs ≥ 100 noncardiac surgeries per month, and if anesthesia, surgery and hospital leadership agree to manage patients as per the policy being implemented and evaluated in the trial.

Patient-level inclusion criteria:

* Patients >/= 18 years of age undergoing major non-cardiac surgery (a state of hyperfibrinolysis)
* Inpatient surgeries with an estimated >/= 5% risk of RBC transfusion, including open surgeries or laparoscopic surgeries with an estimated duration of >/= 3 hours

Examples of eligible surgeries could include (but are not limited to):

1. General surgery (esophagectomy, gastrectomy, gastric repair, small bowel repair or resection, ostomy formation, colon/rectum repair or resection, colostomy, splenectomy, hepatectomy, pancreatectomy, resection of abdominal mass)
2. Orthopedics (hip fracture repair, pelvic fixation, femur repair / fixation, shoulder / humerus open reduction internal fixation, lower extremity amputation)
3. Spine (vertebrectomy, surgery involving >/= 3 levels)
4. Otolaryngology (glossectomy, mandibulectomy, radical laryngectomy)
5. Thoracic (lung resection or decortication)
6. Vascular (arterial bypass / endarterectomy / aneurysmorrhaphy involving the aorta or proximal vessels off the aorta)
7. Gynecology (hysterectomy)
8. Urology (nephrectomy, cystectomy, prostatectomy, pelvic exenteration)
9. Plastic surgery (large neoplasm resections, burns or debridements)
10. Surgeries anticipated to be associated with 5% or greater risk of RBC transfusion in hospital as per the surgical team.

Exclusion Criteria:

* Active thromboembolic disease (i.e., arterial or venous thrombosis within 90 days preoperative)
* Pregnancy
* Cardiac surgery and hip and knee arthroplasty where TXA is standard-of-care
* Surgeries with free flap reconstruction
* Trauma surgeries where TXA was administered within the previous 3 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8421 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients transfused RBCs | From date of surgery until the date of hospital discharge, assessed up to 90 days
  Proportion of patients requiring transfused RBCs
Incidence of DVT or PE (collectively called venous thromboembolism (VTE) | Within 90 days of surgery
  Number of patients with VTE events

SECONDARY OUTCOMES:
Transfused units | From date of surgery until 3 days post-operative, 7 days post-operative, and until the date of hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  The number of RBC units transfused (both at hospital level and patient level).
Arterial event - myocardial infarction | Hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  Secondary safety outcomes include the in-hospital diagnosis of myocardial infarction
Arterial event - stroke | Hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  Secondary safety outcomes include the in-hospital diagnosis of stroke
Venous thrombotic event - deep vein thrombosis | Hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  Secondary safety outcomes include the in-hospital diagnosis of deep vein thrombosis
Venous thrombotic event - pulmonary embolus | Hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  Secondary safety outcomes include the in-hospital diagnosis of pulmonary embolus
Length of hospitalization | Length of index hospital admission
  Hospital length of stay
Intensive care unit (ICU) admission | Hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  Proportion of participants requiring ICU admission
Hospital survival | Hospital discharge. The estimated mean hospital length of stay is anticipated to be <7 days.
  Proportion of patients alive at hospital discharge
90 day survival | Up to day 30
  Survival at 90-days post-operative
Compliance | Intraoperative
  The proportion of enrolled patients who receive a minimum of one dose of the study intervention
Clinical -a patient centered outcome | Up to day 30 postoperative
  Number of days alive and out of hospital 30 (a patient-centered outcome, that integrates length of stay, readmission and early deaths after surgery into a single outcome metric

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Zarychanski, MD, Principal Investigator — University of Manitoba
Locations (10):
- Canada (10):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - University of Manitoba- HSC Campus, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Health Sciences North Research Institute, Greater Sudbury, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute- General Campus, Ottawa, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - Ottawa Hospital Research Institute- Civic Campus, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data to other researchers.

REFERENCES:
- [Derived] Houston BL, McIsaac DI, Breau RH, Andrews M, Avramescu S, Bagry H, Balshaw RF, Daya J, Duncan K, Harle C, Jacobsohn E, Kerelska T, McIsaac S, Ramsay T, Saha T, Perelman I, Recio A, Solvason D, Szoke D, Tenenbein M, Fergusson DA, Zarychanski R. Hospital policy of tranexamic acid to reduce transfusion in major non-cardiac surgery (TRACTION): protocol for a phase IV randomised controlled trial. BMJ Open. 2024 Jun 3;14(6):e084847. doi: 10.1136/bmjopen-2024-084847. PMID 38830735